CLINICAL TRIAL: NCT02052583
Title: Evaluation de l'oxymétrie cérébrale à Deux Niveaux d'Hypothermie thérapeutique après arrêt Cardiaque Extra-hospitalier
Brief Title: Cardiac ARrest : Brain OXymetry Depending on HYpothermia Depth
Acronym: CARBOXHYD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-AOI-02; 2013-A01192-43 (Other: ANSM)
Record Dates: First submitted 2013-11-20; First posted 2014-02-03 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Oxymetry; Hypothermia
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 34°C (Experimental): therapeutic hypothermia at 34 ° C
  Interventions: Procedure: therapeutic hypothermia at 34 ° C
- 32°C (Experimental): therapeutic hypothermia at 32 ° C
  Interventions: Procedure: therapeutic hypothermia at 32 ° C

INTERVENTIONS:
Procedure: therapeutic hypothermia at 32 ° C
  Arms: 32°C
Procedure: therapeutic hypothermia at 34 ° C
  Arms: 34°C

SUMMARY:
Cardiac arrest is a major public health problem, with 700 000 cases per year , and a survival ranging from 4 to 33%. The post- anoxic encephalopathy remains the most serious complication with only a third of survivors . It is due to a series of phenomena involving microcirculation disorders . Cerebral oximetry is a new technique to evaluate the microcirculatory status . To this day it is used in cardiovascular surgery at risk of cerebral hypoperfusion where desaturation of cerebral oximetry is synonymous with ischemia and microcirculatory disorders. Therapeutic hypothermia is the only treatment improves the outcome of patients after extra- hospital cardiac arrest resuscitation . Its mechanisms of action seem to change all the phenomena responsible for microcirculatory reperfusion disorders . Currently it is recommended to practice hypothermia between 32 and 34 ° C. However, a recent study suggests a superiority of hypothermia at 32 ° C rather than 34 ° C.

The hypothesis of this study is that cerebral oximetry value will be different in patients subjected to two different levels of therapeutic hypothermia in the aftermath of an extra- hospital cardiac arrest. These data allow a better understanding of the mechanisms underlying the benefit of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with an extra-hospital cardiac arrest resuscitation and to benefit from therapeutic hypothermia using a servo system to its temperature (CoolGard 3000 ® system)
* Age> 18 years and <80 years

Exclusion Criteria:

* Major Patient protected by law
* Private person administrative or judicial freedom
* Neurological or traumatic cause of cardiac arrest
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Mesure of cerebral oximetry | 8 times during the first 48 hours of hospitalization
  During the first 48 hours of hospitalization, we will collect the cerebral oximetry values in the two cerebral hemispheres.

SECONDARY OUTCOMES:
The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome. | 8 times during the first 48 hours of hospitalization
  The cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor neurological outcome.
For each level of therapeutic hypothermia the cerebral oximetry values will be compared between patients with good and poor becoming | baseline, when target temperature is reached, 6 hours, 12 hours, 18 hours, 24 hours, when 37°C is reached
  For each level of therapeutic hypothermia (32 or 34 ° C), the cerebral oximetry values (average of the two hemispheres) will be compared between patients with good and poor becoming according to the CPC score (CPC = 1 become good score - 2 and bad become CPC = 3-5).
Outcome of patients | 6 months after hospitalization
  The outcome of patients (score 1-2 vs. CPC. 3-5 CPC) will be compared with the level of hypothermia (32 or 34 ° C)
Mesure of lactate | 4 times during the first 48 hours of hospitalization
  Lactate will be compared between patients with good (CPC 1-2) and poor (CPC 3-5) become throughout the study population

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ORBAN, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CH de Fréjus-Saint Raphael, Fréjus
  - CHU de Nice - Hôpital Saint Roch, Nice